CLINICAL TRIAL: NCT06934291
Title: Clinical and Patient-Centered Outcomes of Full-Mouth Ultrasonic Debridement for Periodontitis: A Randomized Controlled Trial Comparing Piezoelectric and Magnetostrictive Devices
Brief Title: Full Mouth Ultrasonic Debridement Carried Out With Either Piezoelectric or Magnetostrictive Device
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Nicola Discepoli, Associate Professor, University of Siena
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MP001
Record Dates: First submitted 2025-03-31; First posted 2025-04-18 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Periodontitis, Adult
Keywords: periodontitis; patient centred outcomes; magnetostrictive
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis | interventions — Emergency Treatment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Piezoelectric (Active Comparator): Full-mouth ultrasonic debridement will be performed with a ultrasonic tip (vibration frequence >18 kHz) powered by a piezoelectric device
  Interventions: Device: Full-mouth ultrasonic debridement with piezoelectric device (EMS, mini piezon)
- Magnetostrictive (Experimental): Full-mouth ultrasonic debridement will be performed with a ultrasonic tip (vibration frequence >18 kHz) powered by a magnetostrictive device.
  Interventions: Device: Full-mouth ultrasonic debridement with magnetostrictive device (Cavitron Select, Dentsply)

INTERVENTIONS:
Device: Full-mouth ultrasonic debridement with piezoelectric device (EMS, mini piezon) — the use of ultrasonic oscillating tips allows supragingival and subgingival biofilm and dental calculus removal
  Arms: Piezoelectric
Device: Full-mouth ultrasonic debridement with magnetostrictive device (Cavitron Select, Dentsply) — the use of ultrasonic oscillating tips allows supragingival and subgingival biofilm and dental calculus removal
  Arms: Magnetostrictive

SUMMARY:
The treatment of periodontitis requires the removal of dental biofilm through both professional mechanical plaque removal and at-home oral hygiene practices. This study aims to compare clinical and psychological outcomes following professional treatment using either piezoelectric or magnetostrictive ultrasonic devices.

DETAILED DESCRIPTION:
Patients diagnosed with periodontitis will be screened for eligibility criteria. A comprehensive full-mouth periodontal assessment will be conducted by a calibrated examiner to determine the severity and extent of the disease. Subsequently, patients will receive oral hygiene instructions, and group allocation will be revealed using a sealed envelope. Based on the assigned group, full-mouth ultrasonic debridement will be performed by a trained operator. Patient perceptions regarding the treatment will then be recorded. After three months, patients will return for a follow-up periodontal evaluation.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* periodontitis of stage 1 and 2
* absence of systemic chronic disease

Exclusion Criteria:

* anticoagulants treatment
* antibiotic treatment 3 months before the screening visit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Pain perception | through study completition, on average 6 months
  vas scale (0-10) for perception of pain after treatment
noise | through study completition, on average 6 months
  vas scale (0-10) for perception of noise after treatment
vibration | through study completition, on average 6 months
  vas scale (0-10) for perception of vibration after treatment

SECONDARY OUTCOMES:
pocket closure | through study completition, on average 6 months
  change of pocket probing depth (millimeter) after treatment measured with a periodontal probe

CONTACTS AND LOCATIONS:
Locations (1):
- AOUS, Siena, SI, Italy

IPD SHARING:
Plan to Share IPD: No